CLINICAL TRIAL: NCT06465043
Title: HFPEF-project: Heart Failure Phenotyping - Exploring the Fingerprints Prospective Observational Study Aiming At Detailed Characterization and Deep Phenotyping of Patients with Heart Failure and Preserved Ejection Fraction (LVEF>40%)
Brief Title: HFPEF-project: Heart Failure Phenotyping - Exploring the Fingerprints
Status: Recruiting | Type: Observational
Sponsor: University of Helsinki (Other)
Collaborators: Aarne Koskelo Foundation (Other); Finnish Foundation for Cardiovascular Research (Other)
Responsible Party: Principal Investigator, Johan Lassus, Principal Investigator, University of Helsinki
Other Study IDs: HUS/628/2024
Record Dates: First submitted 2024-05-09; First posted 2024-06-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-09

CONDITIONS: Heart Failure with Preserved Ejection Fraction
Keywords: HFpEF; iCPET; heart failure; invasive hemodynamics
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine, Stools
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
With an ageing population, the number of patients with heart failure with preserved ejection fraction (HFpEF) or diastolic heart failure is increasing rapidly. This condition is associated with significantly increased morbidity and mortality, but effective treatment options that improve prognosis are very limited.

Further understanding of the nature and determinants of this disease is needed to develop better treatments of HFpEF and to improve the prognosis and quality of life of these patients.

This study will collect a comprehensive, prospective dataset of patients with HFpEF and determine which factors influence the prognosis of this patient group.

The specific aim is to create an accurate description of the spectrum and subtypes of HFpEF enabling better tools to plan and implement individualised treatment for patients.

The main objectives of the study are:

* to describe and categorize the phenotype of HFpEF patients (deep phenotyping) using the latest biochemical, functional and imaging techniques
* identifying factors affecting prognosis and potential new prognostic markers
* prospective follow-up of a contemproary cohort of HFpEF patients to assess outcomes, such as hospitalisations for heart failure, mortality, and quality of life
* identification of specific or aberrant HFpEF phenotypes for genetic studies.

Target population:

* Patients (minimum18 years old) with hospitalization for heart failure (1' or 2' cause for hospitalization) or outpatients with heart failure AND
* Left ventricular ejection fraction (LVEF) >40% within 12 months prior to or during index hospitalization (assessed by ECHO, MRI, LV-cineangiography or radionuclide imaging) AND
* Elevated BNP/NTproBNP AND
* Impaired myocardial relaxation (diastolic dysfunction) assessed by tissue doppler imaging (TDI) velocities on ECHO: lateral mitral annulus velocity (lat E') >9cm/s or septal annulus velocity (sept E') >8 cm/s
* Both de-novo HF and patients with previously diagnosed HF will be eligible

The study prospective, observational study is carried out at Helsinki and Uusimaa Hospital District (HUS).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalisation for heart failure or debilitating dyspnoea (NYHA II-IV) and a diagnosis of HFpEF.
* Left ventricular ejection fraction (LVEF) >40% in the preceding 12 months or during a period of hospitalisation as determined by either cardiac ultrasound, MRI, left ventricular echocardiography, or isotope imaging.
* NTproBNP > 300 pg/ml (or BNP > 100 pg/ml) during hospitalisation or NTproBNP > 125 pg/ml in outpatients.
* Impaired myocardial relaxation (diastolic dysfunction) as determined by tissue doppler imaging (TDI: lateral mitral annulus velocity, lat E' <9cm/s or septal annulus velocity, sept E' <8 cm/s)
* Both previously undiagnosed, de-novo heart failure patients and patients admitted to hospital for acute exacerbation of known heart failure will be included in the study.

Exclusion Criteria:

* Age >85 years
* Significant aortic valve stenosis (AVA ≤1.0 cm2)
* Primary (structural) mitral valve disease with grade III-IV insufficiency or significant stenosis (MVA<1.5 cm2)
* Other severe valvular defect (e.g. secondary severe mitral or severe tricuspid insufficiency)
* Previous LVEF < 40% (HFrEF or HF with improved EF)
* Recent acute coronary syndrome (< 3 months) or myocardial infarction with ST elevations (STEMI) within 12 months
* Previous open heart surgery (CABG/valvular) or percutaneous valvular interventio
* Previously known specific myocardial disease (hypertrophic cardiomyopathy, non-compaction cardiomyopathy (LVNC), right ventricular arrhythmogenic cardiomyopathy (ARVC), cardiac amyloidosis, cardiac sarcoidosis, haemochromatosis)
* End-stage renal disease (eGFR <15 ml/min or dialysis treatment, previous kidney transplantation)
* Significant physical disability, mobility limitation, or dependence on another person for assistance (patient is not self-sufficient) limits participation in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HFpEF hospitalised or attending cardiology outpatient clinic at Helsinki and Uusimaa Hospital District
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
All- cause mortality | 1 year
  Death from any cause

SECONDARY OUTCOMES:
Heart Failure Hospitalisation | 12 months
  Rate of hospitalisation for worsening heart failure
All cause mortality | 5 years
  Death from any cause
Cardiovascular mortality | 1 year
  Death from cardiovascular causes

OTHER OUTCOMES:
Functional status | 6 months
  6-minute walking test (walk distance in meters)

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: Undecided